CLINICAL TRIAL: NCT07338955
Title: Validating and Assessing Reliability of the Urdu Version of the Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire.
Brief Title: Validating and Assessing Reliability
Status: Recruiting | Type: Observational
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Rabia Khan, Assistant Professor, Bahria University
Other Study IDs: BUHS-ERC#001\DPT\25
Record Dates: First submitted 2025-12-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Upper Limb Disability
Keywords: Validation and Reliability of DASH Questionnaire
MeSH Terms: interventions — ethinyl estradiol, levonorgestrel drug combination; Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 385 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Data will be collected from experienced physiotherpist
  Interventions: Other: All participants (Aviane); Other: data collection

INTERVENTIONS:
Other: All participants (Aviane) — Data will be collected from patients having upper limb pain or disability
Other: data collection — Data will be collected from patients having upper limb pain or disbility

SUMMARY:
This study aims to translate, culturally adapt, and validate the Urdu version of the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire for individuals with upper limb disabilities. Since no validated Urdu version currently exists, Urdu-speaking patients face communication barriers that may lead to inaccurate assessment and limited clinical decision-making. By ensuring semantic equivalence through forward-backward translation and expert review, the study seeks to develop a version that is both linguistically accurate and culturally appropriate.

DETAILED DESCRIPTION:
This study aims to translate, culturally adapt, and validate the Urdu version of the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire for individuals with upper limb disabilities. Since no validated Urdu version currently exists, Urdu-speaking patients face communication barriers that may lead to inaccurate assessment and limited clinical decision-making. By ensuring semantic equivalence through forward-backward translation and expert review, the study seeks to develop a version that is both linguistically accurate and culturally appropriate.

A cross-sectional research design will be used, involving adults aged 18-45 years diagnosed with upper limb functional limitations. Participants will complete both the Urdu and English DASH questionnaires to evaluate reliability and validity. Reliability will be assessed through internal consistency (Cronbach's alpha) and test-retest stability (ICC), while validity will be examined using expert scoring (CVI) and correlation with the original instrument. Data analysis will follow standard psychometric testing procedures using SPSS.

The expected outcome is a reliable, valid tool for assessing upper extremity disability in Urdu-speaking populations. This will improve clinical assessment, enhance patient communication, and support broader inclusion in rehabilitation research and practice.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with any upper limb disability or deformity . Able to read, understand and speak Urdu. Individuals with symptoms enduring for at least one week .

Exclusion Criteria:

Cognitive impairment or psychiatric illness that hinders understanding of the questionnaire.

Patients with congenital deformities. Refusal to give informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with upper limb disability or pain for more than 4 weeks
Sampling Method: Non-Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
reliability and validity | December 2025 to January 2026
  To assess the reliability and validity of the Urdu version of the DASH Questionnaire.

SECONDARY OUTCOMES:
cultural adaptation | October 2025 to November2025
  To ensure the cultural adaptation, response of the patient and to compare the results of DASH Questionnaire Urdu version with English version of DASH Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Basakci Calik B, Demir P, Gur Kabul E, Caglayan BC, Keskin A, Karasu U. Validity and Reliability of the Turkish Version of the DASH-TR Questionnaire in Rheumatoid Arthritis Patients, Based on Rasch Analysis. Int J Rheum Dis. 2022 Aug;25(8):851-860. doi: 10.1111/1756-185X.14358. Epub 2022 Jun 6. PMID 35665605
- [Result] Puentes Gutierrez AB, Garcia Bascones M, Jimenez Diaz F, Cuena Boy R, Puentes Gutierrez R. [Validity and reliability of DASH questionnaire in women who suffer from lymphedema as a side effect of a breast cancer treatment]. Rehabilitacion (Madr). 2023 Jul-Sep;57(3):100780. doi: 10.1016/j.rh.2022.100780. Epub 2023 Feb 3. Spanish. PMID 36739630